CLINICAL TRIAL: NCT03762551
Title: Expression of Janus Kinase 1 in Vitiligo and Psoriasis Before and After Narrow Band UVB: a Case-Control Study
Brief Title: Janus Kinase 1 in Vitiligo & Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dermatology 11
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2015-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitiligo (Experimental): assess the level of JAK1 in vitiligo patients before and after treatment with NB-UVB
  Interventions: Other: skin biopsy
- psoriasis (Active Comparator): assess the level of JAK1 in psoriasis patients before and after treatment with NB-UVB
  Interventions: Other: skin biopsy
- controls (Other): assess the level of JAK1 in controls
  Interventions: Other: skin biopsy

INTERVENTIONS:
Other: skin biopsy — Two (4 mm) punch skin biopsies were taken from the 20 patients; one prior to the initiation of phototherapy and the other after the last session (from the same site). One skin biopsy was taken from the skin of each of the 10 control healthy participants. Skin biopsy specimens were preserved in Radio-Immunoprecipitation Assay (RIBA) buffer.

SUMMARY:
Assessment of the level of JAK1 in both vitiligo and psoriasis patients before and after treatment with NB-UVB which is considered a gold standard therapy for both diseases.

ELIGIBILITY:
Inclusion Criteria:

* age above 12 years of age.
* psoriasis vulgaris or non-segmental vitiligo
* patients who received no systemic or topical treatment at least 6 weeks prior to enrollment into the study.

Exclusion Criteria:

* psoriasis patients with erythrodermic psoriasis, pustular psoriasis or associated psoriatic arthritis
* vitiligo patients with segmental or universal vitiligo were excluded from the study.
* any patient with a photosensitive disorder or any contraindication to phototherapy exposure, e.g., history or presence of malignant or premalignant skin lesions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the tissue level of JAK1 in both vitiligo and psoriasis patients before and after treatment with NB-UVB | 1 year